CLINICAL TRIAL: NCT06022835
Title: Tegaderm(TM) Chlorhexidine Gluconate-gel (CHG) Dressing for the Prevention of Exit Site Infection in Patients Receiving Peritoneal Dialysis.
Brief Title: Chlorhexidine Gluconate-gel Dressing for Exit Site Infection in Peritoneal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group, Singapore (Other Government)
Responsible Party: Principal Investigator, Allen Liu Yan Lun, Senior Consultant, National Healthcare Group, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019/00493
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Peritoneal Dialysis Catheter Exit Site Infection; End Stage Renal Disease on Dialysis; Dialysis; Complications
Keywords: peritoneal dialysis; exit site infection; chlorhexidine; dressing; End stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Chromogranins; Bandages

STUDY DESIGN:
Intervention Model Description: The recruitment period was from October 2019 to August 2022. All incident PD patients aged between 21-99 years were screened. Patients allergic to chlorhexidine and Tegaderm dressing were excluded from the study. One hundred thirty-eight patients initiated PD and were screened between October 2019 and April 2022.
  A historical cohort of incident PD patients from November 2016 to October 2017 with the same inclusion and exclusion criteria were also recruited and compared to the CHG dressing group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chlorhexidine Gluconate-gel (CHG) Dressing group (Experimental): Participants used Tegaderm™ CHG dressing for 4 months. The dressing was changed every seven days or soiled.
  Interventions: Other: Chlorhexidine Gluconate-gel (CHG) Dressing

INTERVENTIONS:
Other: Chlorhexidine Gluconate-gel (CHG) Dressing — Participants used Tegaderm™ CHG dressing for 4 months. The dressing was changed every seven days or soiled.

SUMMARY:
Exit site infection (ESI) is one of the major predisposing factors to peritoneal dialysis (PD) related peritonitis. Chlorhexidine Gluconate (CHG) has been widely used for cutaneous disinfection for half a century. TegadermTM CHG is a water-proof dressing with gel pads that provide 2% CHG to the skin surface and effectively prevents catheter-related infections for intravascular catheters. However, its use has not been accessed in patients with PD catheters. We aim to evaluate the effectiveness of TegadermTM CHG dressing in preventing ESI in PD patients.

DETAILED DESCRIPTION:
Peritoneal Dialysis (PD) is one of the common therapies for patients with End Stage Renal Failure (ESRF). As the global burden of chronic kidney disease continues to increase, so does the need for a cost-effective renal replacement therapy (1). Patient outcomes with peritoneal dialysis are comparable to or better than those with haemodialysis, and peritoneal dialysis is also more cost-effective (1). It is reported that PD improves patient's well-being and has greater personal freedom as compared to Hemodialysis through less restrictive life-style changes (2). All dialysis treatments include a certain risk of infection because of the decreased immune defenses of patients in established renal failure (ERF) and because dialysis techniques increase the potential of microbial contamination (3).

PD is associated with a high risk of infection of the peritoneum, subcutaneous tunnel and catheter exit site (4). ESI is diagnosed by the presence of purulent drainage, with or without erythema of the skin at the catheter-epidermal interface (5). Exit site infection (ESI) increases the possibility of developing PD peritonitis which demands careful attendance to these problems. It is estimated that 12% of cases of ESI results in PD peritonitis (6). As many as 15%-50% of ESRF patients are on PD, but recurrent or prolonged peritonitis may causes technique failure in PD (3). The majority of catheter related problems are of an infection nature - mainly represented by peritonitis (61%); ESI (23%); catheter obstruction, dislocation and leakage making up the rest (3). Peritonitis can be associated with severe pain leading to hospitalisation, catheter loss, and a risk of death; and it therefore continues to be a serious complication for PD patients (7).

There are no recommendations what topical care of the PD catheter exit site is optimal. Several methods including Povidone-Iodine, hydrogen peroxide, chlorhexidine, soap and water, and topical creams such as gentamicin or mupirocin cream have been studied for exit site care (8,9).

A number of topical cleansing agents have been studied for prevention of catheter-related infections however no cleansing agent has shown to be superior with respect to preventing catheter-related infections (5). The International Society for Peritoneal Dialysis (ISPD) recommends the use of daily topical application of antibiotic cream or ointment to the catheter exit site to prevent infection and exit site be cleansed at least twice weekly and every time after a shower (5).

Appropriate care of the exit site will avoid loss of catheter and unnecessary dialysis modality change. PD-related infection is the most common cause of technique failure. Prevention and treatment of PD catheter related infection such as peritonitis and exit site infections are important to maintain on PD therapy.

In Khoo Teck Puat Hospital (KTPH) we had been following the ISPD guidelines on the dressing recommendation to use iodine as the preferred cleansing agent and application of Gentamicin cream 0.1% as prophylaxis to prevent PD exit site infection. However, we had noticed an increase in patient's risk of PD ESI from 2016 0.15/year at risk, 2017 0.19/year at risk and 2018 0.22/year at risk. Of which 40-55% were gram positive infections, 5-15% were gram negative infections and the rest were having no bacterial cultures or fungal infections. We evaluated on the infection episodes and reassessed on patients technique and home environment and found that reasons of infection were due to poor compliance to dressing techniques, frequency of change after shower, hand washing technique and home environment cleanliness.

Several research articles were reviewed and Chlorhexidine Gluconate (CHG) was found to be used widely throughout the world for more than 50 years for cutaneous disinfection, hand hygiene and oral hygiene, and the safety of CHG is well established (10).Clinically relevant high-level bacterial resistance has been very rare (11).

TegadermTM CHG Dressing had a gel pad that provides 2% CHG to the skin surface. It was proven to largely reduce catheter-related bloodstream infections (CRBSI) (from 1.21 to 0.28 per 1000 catheter days) and vascular catheter colonization (12). The CHG dressing is recommended to be worn up to 7days and provide CHG antimicrobial protection, secure adhesion, gentle removal, site visibility, breathability and patient comfort (13).

Unlike CRBSI, TegadermTM CHG Dressing was not evaluated for its effectiveness in prevention of exit infection in PD patients. This would be the first study to evaluate the effectiveness of TegadermTM CHG Dressing in reducing peritoneal dialysis catheter exit site infection. The ease of application of the dressing will help to increase patients and caregivers' compliance as the frequency of change was reduced from daily to once every 7 days. TegadermTM CHG dressing also water-proof and it will helps in maintaining the exit site clean and dry. By reducing the PD ESI rates, it will also helps in preventing secondary peritonitis and prevents unnecessary dialysis modality changes.

This would be the first study to evaluate the effectiveness of Tegaderm™ chlorhexidine gluconate-gel (CHG) dressing for the prevention of exit site infection in patient receiving peritoneal dialysis.

Participants will use Tegaderm™ chlorhexidine gluconate-gel (CHG) dressing for a period of 4-6months. Results will be compared with historical data from 1st Nov 2016 to 31st Oct 2017. Estimated 40 patient's historical data will be reviewed.

New Method:

Patients are taught to perform 7 steps handwashing, clean PD exit site with chlorhexidine swab sticks, dry with gauze, and apply TegadermTM CHG Dressing. This has to be repeated every 7days or when the dressing is soiled.

Old Method:

Patients are taught to perform 7 steps handwashing, clean PD exit site with 3 swab sticks, dry with gauze, apply Gentamicin cream 0.1% and cover with soft cloth dressing. This has to be repeated daily after shower or when the dressing is soiled.

References

1. Kam TL, Chow KM, Luijtaarden M, Johnson DW, Jager KJ, Mehrotra, JR, Naicker, S, Pecoits-Filho R, Yu XQ, Lameire N: Changes in the worldwide epidemiology of peritoneal dialysis. Nature Reviews Nephrology, 13:90-109-3, 2017
2. Lockwood C, Hodgkinson B, Page T: Clinical effectiveness of different approaches to peritoneal dialysis catheter exit-site care. JBI Reports, 1(6): 167-201, 2003
3. Akoh JA: Peritoneal dialysis associated infections: An update on diagnosis and management. World Journal of Nephrology, 1(4):106-122, 2012
4. Bianchi P, Buoncristiani E, Buoncristiani U: Antisepsis. Contrib Nephrol 154: 1-6, 2007
5. Szeto CC, Kam TL, Johnson DW, Bernardini J, Dong J, Figueiredo AE, Ito Y, Kazancioglu R, Moraes T, Esch SV, Brown EA: ISPD Catheter-related infection recommendations: 2017 Update. Perit Dial Int, 37: 141-154, 2007
6. Brook NR, White SA, Waller JR, Nicholson ML: The surgical management of peritoneal dialysis catheters. Ann R Coll Surg Engl. 86: 190-195. 2004
7. Campos RP, Chula DC, Riella MC: Complications of the peritoneal access and their management. Contrib Nephrol, 163: 183-197, 2009
8. Ques AAM, Campo MV, Arribas CM, Marcos BB, Ramos CQ, del Barrio OR, Cortes MP, Marenco MT: Effectiveness of different types of care for the peritoneal dialysis catheter exit site: A systematic review. JBI Database of Systematic Reviews and Implementation Reports, 11(9):133-179, 2013
9. McCormack K, Rabindranath K, Kilonzo M, Vale L, Fraser C, Mclntyre L, Thomas S, Rothnie H, Fluck N, Gould IM, Waugh N: Systematic review of the effectiveness of preventing and treating Staphylococcus aureus carriage in reducing peritoneal catheter-related infections. Health Technol Assess, 11(23):iii-iv, ix-x, 1-66, 2007
10. Milstone AM. Passaretti CL. Perl TM. Chlorhexidine: expanding the armamentarium for infection control and prevention. Clin Infec Dis. 46:274-81, 2008
11. McDonnell G, Russell AD. Antiseptics and disinfectants: activity, action, and resistance. Clin Microbiol Rev, 12(1): 147-79, 1999
12. Righetti M, Palmieri N, Bracchi O, Prencipe M, Bruschetta E, Colombo F, et al.: Tegaderm CHG dressing significantly improves catheter-related infection rate in hemodialysis patients. The journal of vascular access, 17(5):417-22, 2016
13. https://multimedia.3m.com/mws/media/501550O/tegaderm-chg-dressing-product-brochure.pdf

ELIGIBILITY:
Inclusion Criteria:

All incident PD patients

Exclusion Criteria:

Patients allergic to chlorhexidine and Tegaderm dressing

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
The incidence rate of exit site infection | 12 weeks
  the rate in patient months and by percentage

SECONDARY OUTCOMES:
time to first ESI and PD-associated peritonitis | 12 weeks
  Number of days patients have ESI/peritonitis-free survival
PD-associated peritonitis | 12 weeks
  based on ISPD guidelines
PD-related hospitalisation rate | 12 weeks
  hospitalisation rate in patient months

CONTACTS AND LOCATIONS:
Overall Officials: Allen Yan Lun Liu, Study Chair — Khoo Teck Puat Hospital, Singapore
Locations (1):
- Allen Liu, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No